CLINICAL TRIAL: NCT04236973
Title: Multicentre Clinical Performance Evaluation of the Molbio Diagnostics Truenat™ HCV RNA Assay
Brief Title: Truenat™ HCV RNA Assay Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: HC014
Record Dates: First submitted 2020-01-15; First posted 2020-01-22 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- clinical performance of the Truenat™ HCV assay (Experimental): The study will be conducted in different geographical regions and populations and is designed to meet requirements of the Common Technical Specifications 2009/886/EC (CTS) of the CE-IVDD and WHO TSS-10 (draft) for IVDs medical devices used for the qualitative and quantitative detection of Hepatitis C RNA.
  Interventions: Device: Molbio Truenat™ HCV assay (the investigational product)
- comparison CE-IVD marked reference assay arm (Active Comparator): Plasma specimens from the participants will be tested on Abbott RealTime HCV assay that is approved for HCV diagnostics use by countries' authorities.
  Interventions: Other: Abbott RealTime HCV assay

INTERVENTIONS:
Device: Molbio Truenat™ HCV assay (the investigational product) — The Molbio Truenat™ HCV assay (the investigational product) is a quantitative chip-based Real Time Reverse Transcription Polymerase Chain Reaction (qRT-PCR) tests for the detection of HCV genomic RNA from human whole blood, EDTA plasma and serum. The Truenat™ HCV assay runs on the Truelab™ Uno, Truelab™ Duo or Truelab™ Quadro Dx. Results of testing by Truenat™ HCV assay will not be used to make any clinical decisions, and should not be communicated to study participants.
  Arms: clinical performance of the Truenat™ HCV assay
Other: Abbott RealTime HCV assay — Plasma specimens will be also tested on Abbott RealTime HCV assay that is approved for HCV diagnostics use by countries' authorities. Only the results of Abbott RealTime HCV assay may be used to make clinical decisions.
  Arms: comparison CE-IVD marked reference assay arm

SUMMARY:
Molbio Diagnostics Ltd. (India) has developed the Truelab™ Real Time quantitative PCR system that is widely used in India for diagnostics of tuberculosis (TB). The system consists of two portable machines and two microfluidic cartridges and can be used in point-of-care settings. The manufacturer has recently developed a new assay that detects HCV RNA, the Truenat™ HCV RNA assay. It is a simple two-step assay for RNA extraction and amplification with a total turnaround time of 60 min, using whole blood, plasma and serum as sample types. Most importantly, the assay can be performed from a drop of capillary blood eliminating the need for venous access and blood draw and increasing its usability in the settings where phlebotomy service are not available. To date, validation of the assay was performed using archived plasma specimens and contrived whole blood specimens. FIND aims to conduct a multicentre evaluation to assess the assay's sensitivity, specificity and quantitative accuracy in freshly collected whole blood, plasma and serum specimens from target populations. The evaluation aims to gather performance data in line with the requirements set forth in the Common Technical Specifications 2009/886/EC (CTS) of the CE In Vitro Diagnostics Medical Devices Directive 98/79/CE (CE-IVDD), as well as the World Health Organization (WHO) Technical Specification Series 10 (draft) (TSS-10) for In vitro diagnostic (IVDs) medical devices used for the qualitative and quantitative detection of HCV RNA.

DETAILED DESCRIPTION:
Even though hepatitis C virus (HCV) infection can now be cured, globally, fewer than 20% of the 71 million living with HCV are aware of their status; diagnosis remains a major challenge. While serology screening tests that detect the presence of antibodies against HCV, can be performed in decentralized settings, these tests cannot distinguish between resolved (about 25% of seropositive cases) and active infection. Therefore, positive serology test results require further confirmation by laboratory-based methods that detects the viral particle. The two-step testing process results in high drop-off in confirmatory testing among HCV seropositive individuals, especially in low- and middle-income countries (LMIC) where laboratory infrastructure is lacking. Providing access to confirmatory testing in decentralized settings has a high potential to increase the coverage of HCV testing services in LMIC.

Molbio Diagnostics Ltd. (India) has developed the Truelab™ Real Time quantitative PCR system that is widely used in India for diagnostics of tuberculosis (TB). The system consists of two portable machines and two microfluidic cartridges and can be used in point-of-care settings. The manufacturer has recently developed a new assay that detects HCV RNA, the Truenat™ HCV RNA assay. It is a simple two-step assay for RNA extraction and amplification with a total turnaround time of 60 min, using whole blood, plasma and serum as sample types. Most importantly, the assay can be performed from a drop of capillary blood eliminating the need for venous access and blood draw and increasing its usability in the settings where phlebotomy service are not available. To date, validation of the assay was performed using archived plasma specimens and contrived whole blood specimens. FIND aims to conduct a multicentre evaluation to assess the assay's sensitivity, specificity and quantitative accuracy in freshly collected whole blood, plasma and serum specimens from target populations. The evaluation aims to gather performance data in line with the requirements set forth in the Common Technical Specifications 2009/886/EC (CTS) of the CE In Vitro Diagnostics Medical Devices Directive 98/79/CE (CE-IVDD), as well as the World Health Organization (WHO) Technical Specification Series 10 (draft) (TSS-10) for In vitro diagnostic (IVDs) medical devices used for the qualitative and quantitative detection of HCV RNA. The data will be published as a peer-reviewed report and made available to the test manufacturer to support regulatory submissions.

ELIGIBILITY:
Inclusion Criteria:

Individuals reached the age of an adult as defined in the country that are able to understand the scope of the study and provide informed consent will be invited to take part in the study. In order to meet the study objectives, four different population groups will be considered:

1. HCV SEROPOS: Individuals at risk of having HCV infection based on positive HCV serology test results, without history of HCV treatment

   Inclusion criterion:

   • Documented positive result of HCV serology test
2. HCV RISK: Individuals with unknown serology status at risk of HCV infection based on past and/or current exposure to risk factors

   Inclusion criterion:

   • Past and/or current exposure to one of the high risk factors as defined by WHO and CDC guidelines (Appendix 1)
3. HCV TREAT: Individuals diagnosed with chronic HCV infection who initiated or completed the anti-HCV treatment with direct acting antivirals (DAA) presenting at the clinical site for treatment monitoring or test of cure (i.e. sustained virological response)

   Inclusion criterion:

   • Initiated on DAA treatment (regardless of type of DAA regimen) within 12 months prior to the enrolment to the study
4. BLOOD DONORS: Healthy blood donors free of HBV, HCV and HIV infections, as determined by standard blood bank protocols

Exclusion Criteria:

Exclusion criteria (for all study populations):

* Previously enrolled in the study
* Unwilling or unable to provide required volume of fingerstick blood
* Unwilling or unable to provide required volume of venous whole blood

Exclusion criterion for BLOOD DONORS:

• Positive results in HBV, HCV and HIV tests routinely used in the blood bank to assess blood products safety

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1330 (Actual)
Dates: Start 2020-01-12 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Point estimates of clinical sensitivity and specificity | From day 1 (enrolment) up to day 30 (completion of the reference testing)
  Point estimates (with 95% confidence intervals) of clinical sensitivity and clinical specificity of the Truenat™ HCV assay in fingerstick blood and plasma measured against Abbott RealTime HCV assay in plasma. Sensitivity and specificity of the Truenat™ HCV assay will be obtained for each sample type separately, using Abbott RealTime HCV assay as a reference method.
Accuracy of quantification of HCV viral load level in fingerstick blood and plasma by the Truenat™ HCV assay | From day 1 (enrolment) up to day 30 (completion of the reference testing)
  To evaluate the quantitative performance of the Truenat™ HCV assay in fingerstick blood and plasma specimens, assay results for each specimen type within the linear range will be compared with the results of Abbott RealTime HCV assay performed from a paired plasma specimen. The data will be visualized with the use of scatter plots, and analyzed using Deming regression. The resulting slope of the regression fir will be reported, with 95% confidence intervals.
  In addition to the linear regression analysis, a Bland-Altman plot will also be generated.
  The percentage of samples with results >0.5 Log IU/mL apart in quantitation between the test and the reference method will be reported.

SECONDARY OUTCOMES:
Level of agreement between result outputs of the Truenat™ HCV assay performed from different specimens. | From day 1 (enrolment) up to day 30 (completion of the reference testing)
  Percentage of agreement between result outputs of the Truenat™ HCV assay performed from different specimen types will be calculated, with 95% confidence intervals based on Wilson's score method, as the percentage of the number of samples with identical results over the total number of samples tested. In addition, the Cohen's k coefficient of agreement will also be calculated as a measure of agreement between different sample types.
Accuracy of quantification of HCV viral load levels in serum and venous whole blood specimens by the Truenat™ HCV assay | From day 1 (enrolment) up to day 30 (completion of the reference testing)
  Evaluation of the correlation of HCV viral load levels determined by the Truenat™ HCV assay in different specimen types, Truenat™ HCV assay results for each specimen type within the linear range will be compared with the results of the same assay in another specimen type. The data will be visualized with the use of scatter plots, and analyzed using Deming regression.
Operational usability of the Truenat HCV assay | From the enrolment of the first participant to the completion of all study procedures for the last enrolled participant and up to 12 months
  Assessment of operational characteristics including but not limited to rate of invalid results, total hands on time, description of operator experience with the assays through the appraisal sheet.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Ivanova, MD, PhD, Study Director — Foundation for Innovative New Diagnostics
Locations (5):
- Aarhus University Hospital, Aarhus, Denmark
- St Paul's Hospital Millennium Medical College, Addis Ababa, Ethiopia
- National Centre for Diseases Control, Tbilisi, Georgia
- HIV-NAT Thai Red Cross AIDS Research Centre, Bangkok, Thailand
- International Charitable Foundation Alliance for Public Health, Kyiv, Ukraine